CLINICAL TRIAL: NCT01584791
Title: Korean Multicenter Randomized Controlled Trial (RCT) of Pidogul for Patients With Coronary Stenting
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Hanmi Pharmaceutical co., ltd. (Other)
Responsible Party: Principal Investigator, Hyo-Soo Kim, Professor, Department of Internal Medicine, Seoul National University Hospital, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KOPIDO STENT
Record Dates: First submitted 2012-04-23; First posted 2012-04-25 (Estimated); Last update posted 2012-04-25 (Estimated); Status verified 2012-04

CONDITIONS: Coronary Artery Disease
Keywords: CAD; PCI; Percutaneous Coronary Intervention
MeSH Terms: conditions — Coronary Artery Disease | interventions — Clopidogrel; Aspirin

ARMS (2):
- clopidogrel napadisilate + aspirin (Experimental)
  Interventions: Drug: clopidogrel napadisilate + aspirin
- clopidogrel bisulfate + aspirin (Active Comparator)
  Interventions: Drug: clopidogrel bisulfate + aspirin

INTERVENTIONS:
Drug: clopidogrel napadisilate + aspirin — clopidogrel napadisilate 75mg + aspirin 100mg
  Arms: clopidogrel napadisilate + aspirin
Drug: clopidogrel bisulfate + aspirin — clopidogrel bisulfate 75mg + aspirin 100mg
  Arms: clopidogrel bisulfate + aspirin

SUMMARY:
The aim of the current study is to compare the antiplatelet efficacy and safety of clopidogrel napadisilate and clopidogrel bisulfate in Coronary Artery Disease (CAD) patients after coronary stent implantation.

ELIGIBILITY:
Inclusion Criteria:

* Korean men and women between the age of 20 and 85
* Patients who were diagnosed as having CAD
* Patients who were planned to undergo PCI

Exclusion Criteria:

* Patients who were not treated with PCI or intended to treat with PCI but failed
* Patients who were were taking or had taken other antiplatelet or anticoagulant for more than 2 weeks within the prior 30 days
* Patients who were had a history of alcohol abuse or intoxication; (4) had hypersensitivity to clopidogrel or aspirin
* Patients who were had hypersensitivity to clopidogrel or aspirin
* Patients who were had abnormal laboratory results indicative of liver disease
* Patients who were had blood coagulation disorders, uncontrolled severe hypertension, active bleeding, or history of severe bleeding, such as intracranial hemorrhage or ulcer bleeding
* Patients who were were pregnant, breastfeeding, or not using effective methods of contraception
* Patients who were had other contraindication to study drug
* Patients who were had participated in another clinical study within 4 weeks prior to the start of this study

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2010-10; Primary Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
The percentage of P2Y12 receptor inhibition | 4 weeks

SECONDARY OUTCOMES:
Adverse events after study medication | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Park JB, Koo BK, Choi WG, Kim SY, Park J, Kwan J, Park CG, Kim HS. Comparison of antiplatelet efficacy and tolerability of clopidogrel napadisilate with clopidogrel bisulfate in coronary artery disease patients after percutaneous coronary intervention: a prospective, multicenter, randomized, open-label, phase IV, noninferiority trial. Clin Ther. 2013 Jan;35(1):28-37.e4. doi: 10.1016/j.clinthera.2012.12.004. PMID 23328268